CLINICAL TRIAL: NCT05749991
Title: A Randomized Controlled Clinical Trial Comparing Fissure Sealant Retention Rate, Chair Time, and Patients' Preference Using Dryshield and Cotton Roll Isolation
Brief Title: Efficacy and Retention of Sealants Placement Using Two Isolation Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuwait University (Other)
Responsible Party: Principal Investigator, ABRAR ALANZI, Associate Professor, Kuwait University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VDR/EC/3344
Record Dates: First submitted 2023-01-23; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Retention; Time; Patient Preference
MeSH Terms: conditions — Patient Preference

STUDY DESIGN:
Intervention Model Description: All eligible study participants were randomised using simple block random allocation to ensure balanced randomization for each isolation system. Each participant was given an envelope and a printed participant number. Each number identified the isolation technique used for sealant placement and the isolation application sequence to be used.
Who Masked: Outcomes Assessor
Masking Description: The participants, care providers and the principle supervisor were not blinded since they know which isolation technique was used during the placement of sealant. But the outcome assessor was blinded and he assessed the sealants placement after 6, 12, and 18 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DryShield Isolation (Experimental): Device: Dryshield DryShield (DS) is an all-in-one isolation system. It combines the tasks of fluid evacuation, tongue and cheek retraction, and serves as a bite block. Its design allows it to suction and isolate half the oral cavity at a time. Dryshield was used to isolate teeth that required sealant placement in the assigned participants.
  Interventions: Device: Dryshield
- Cotton Roll Isolation (Active Comparator): Cotton Roll Isolation requires placing cotton rolls along the buccal mucosa, especially over the parotid glands ducts for maxillary teeth. For the mandibular teeth, the cotton rolls are placed in the buccal vestibule and the floor of the mouth (between the lower buccal mucosa and underneath and/or between the tongue).
  Cotton roll isolation was used to isolate teeth that required sealant placement in the assigned participants.
  With this technique, a high-speed evacuation of saliva and water is used.
  Interventions: Device: Cotton roll isolation

INTERVENTIONS:
Device: Dryshield — DryShield combines the tasks of high-suction evacuator, saliva ejector, bite block, tongue shield, and oral pathway protector in one easy-to-use device.
  The DryShield solution® is a patented autoclavable isolation system (MA, USA)
  Arms: DryShield Isolation
Device: Cotton roll isolation — Cotton Roll Isolation requires placing cotton rolls along the buccal mucosa, especially over the parotid glands ducts for maxillary teeth. For the mandibular teeth, the cotton rolls are placed in the buccal vestibule and the floor of the mouth (between the lower buccal mucosa and underneath and/or between the tongue). With this technique, a high-speed evacuation of saliva and water is used.
  Other Names: Cotton roll
  Arms: Cotton Roll Isolation

SUMMARY:
The trial aimed to evaluate the sealant retention, patient's preference and chair time needed during pit and fissure sealant placement under two isolation techniques [Dryshield system (DS) and cotton roll isolation (CRI)] in a university setting.

DETAILED DESCRIPTION:
In children, 80-90% of dental caries is found in the pits and fissures of the posterior permanent teeth. Pit and fissure sealants (PFS) can be used effectively to prevent dental caries. When applied correctly, dental PFS accomplish three main objectives: preventing dental caries development, hindering dental caries development in its initial phases, and inhibiting the spread of bacteria that cause dental caries. To be effective, PFS need to be applied under sufficient moisture control around the specific teeth undergoing treatment. Therefore, proper isolation of the teeth is one of the most important steps when placing sealants to ensure their retention.

Cotton roll isolation (CRI) has been widely used for sealant placement, and is the most common method among pediatric dentists. However, the placement of cotton rolls on the lateral part of the tongue or inadequate isolation during CRI has both been reported to produce gagging, tasting the contents and requiring frequent replacement of the wet cotton rolls.

A previous study demonstrated that new moisture control systems such as Isolite, produce sealant retention rates comparable to cotton roll isolation, while decreasing procedure time. DryShield (DS) has recently been introduced as an all-in-one isolation system. It is similar to the Isolite as it combines the tasks of fluid evacuation, tongue and cheek retraction, and serves as a bite block, but differs in that it is autoclavable and does not provide illumination. Its design allows it to suction and isolate half the oral cavity at a time. Therefore, it should presumably facilitate sealants placement under a more controlled environment, while reducing chair time for the dentist.

Few trials have compared the PFS chair time and patient acceptance of DS to the CRI. The goals of this study were to evaluate patients' preferences, time efficiency, and retention of PFS using DS compared to CRI in a single randomized clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy patients with no compromising medical or physical condition
2. age ranging from six to 12 years old;
3. patients with at least one caries-free permanent molar in any quadrant, with normal anatomy, who qualified for pit and fissure sealant application with an International Caries Detection and Assessment System (ICDAS) score of 0-2.
4. no prior sealants or restorations on the teeth under study;
5. no cavitated carious lesions;
6. cooperative patients (classified as 3 or 4 according to the Frankl Behavioral Rating Scale)
7. legal guardian consents and approved assents to the child's participation in the study.

Exclusion Criteria:

1. a history of chronic disease (e.g., epilepsy, ectodermal dysplasia, cardiac anomalies);
2. inability to return for follow-ups.
3. patients with molars that have partially erupted
4. a permanent molar with enamel flaws or abnormal anatomy
5. children who are uncooperative, with a Frankl Behaviour Rating Scale of 1 or 2;
6. children who have a severe gagging reflex;
7. special needs children.
8. Those who do not provide appropriate assents or consents

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2018-06-03 (Actual); Primary Completion 2020-02-09 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Change in Fissure Sealant Retention at 6 months | Change in sealant retention at 6 months
  Patients were clinically evaluated by a study supervisor as a blinded outcome assessor after 6 months of sealant placement. The evaluation was according to Simonsen's criteria: Completely retained, Partially retained, or Missing.
Change in Fissure Sealant Retention at 12 months | Change in sealant retention at 12 months
  Patients were clinically evaluated by a study supervisor as a blinded outcome assessor after 12 months of sealant placement. The evaluation was according to Simonsen's criteria: Completely retained, Partially retained, or Missing.
Change in Fissure Sealant Retention at 18 months | Change in sealant retention at 18 months
  assessor after 18 months of sealant placement. The evaluation was according to Simonsen's criteria: Completely retained, Partially retained, or Missing.

SECONDARY OUTCOMES:
Placement time of sealants using Dryshield vs Cotton roll isolation | 0 Day (After the completion of initial sealant placement and removal of the isolation device)
  The placement time for sealant application was recorded with a stopwatch by the dental assistant as follows for the two techniques: the insertion of the isolation aids (DS or CRI) in the oral cavity constituted the start time, and the end time was when the isolation system was completely removed from the participant's mouth after the sealants application.
Patient preference for Dryshield or Cotton roll isolation | 0 Day (After the completion of initial sealant placement and removal of the isolation device)
  A six-item interview-based questionnaire was administered to assess participants' acceptance of the isolation technique used.

CONTACTS AND LOCATIONS:
Overall Officials: Abrar N Alanzi, Principal Investigator — Kuwait University -Faculty of Dentistry
Locations (1):
- Kuwait University Faculty of Dentistry Dental Clinics, Kuwait City, Kuwait

REFERENCES:
- [Background] Ahovuo-Saloranta A, Forss H, Walsh T, Nordblad A, Makela M, Worthington HV. Pit and fissure sealants for preventing dental decay in permanent teeth. Cochrane Database Syst Rev. 2017 Jul 31;7(7):CD001830. doi: 10.1002/14651858.CD001830.pub5. PMID 28759120
- [Background] Jenson L, Budenz AW, Featherstone JD, Ramos-Gomez FJ, Spolsky VW, Young DA. Clinical protocols for caries management by risk assessment. J Calif Dent Assoc. 2007 Oct;35(10):714-23. PMID 18044379
- [Background] Beauchamp J, Caufield PW, Crall JJ, Donly K, Feigal R, Gooch B, Ismail A, Kohn W, Siegal M, Simonsen R; American Dental Association Council on Scientific Affairs. Evidence-based clinical recommendations for the use of pit-and-fissure sealants: a report of the American Dental Association Council on Scientific Affairs. J Am Dent Assoc. 2008 Mar;139(3):257-68. doi: 10.14219/jada.archive.2008.0155. PMID 18310730
- [Background] Straffon LH, Dennison JB, More FG. Three-year evaluation of sealant: effect of isolation on efficacy. J Am Dent Assoc. 1985 May;110(5):714-7. doi: 10.14219/jada.archive.1985.0425. PMID 3159777
- [Background] Primosch RE, Barr ES. Sealant use and placement techniques among pediatric dentists. J Am Dent Assoc. 2001 Oct;132(10):1442-51; quiz 1461. doi: 10.14219/jada.archive.2001.0061. PMID 11680361
- [Result] Collette J, Wilson S, Sullivan D. A study of the Isolite system during sealant placement: efficacy and patient acceptance. Pediatr Dent. 2010 Mar-Apr;32(2):146-50. PMID 20483019
- [Result] Alhareky MS, Mermelstein D, Finkelman M, Alhumaid J, Loo C. Efficiency and patient satisfaction with the Isolite system versus rubber dam for sealant placement in pediatric patients. Pediatr Dent. 2014 Sep-Oct;36(5):400-4. PMID 25303507
- [Result] Mattar RE, Sulimany AM, Binsaleh SS, Al-Majed IM. Comparison of Fissure Sealant Chair Time and Patients' Preference Using Three Different Isolation Techniques. Children (Basel). 2021 May 25;8(6):444. doi: 10.3390/children8060444. PMID 34070253
- [Result] Mattar RE, Sulimany AM, Binsaleh SS, Hamdan HM, Al-Majed IM. Evaluation of fissure sealant retention rates using Isolite in comparison with rubber dam and cotton roll isolation techniques: A randomized clinical trial. Int J Paediatr Dent. 2023 Jan;33(1):12-19. doi: 10.1111/ipd.13008. Epub 2022 May 22. PMID 35543302